CLINICAL TRIAL: NCT01621789
Title: A Descriptive Study to Evaluate the Efficacy of the Dye Compound of the Combination of Lutein, Zeaxanthin and Trypan Blue to Stain the Anterior Lens Capsule During Cataract Phacoemulsification.
Brief Title: Efficacy of Lutein, Zeaxanthine and Trypan Blue to Stain the Anterior Lens Capsule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rubens Belfort Jr., Full Professor of Ophthalmology, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CEP 2146/11
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Cataract
Keywords: lutein; zeaxanthin; trypan blue; dye
MeSH Terms: conditions — Cataract | interventions — Zeaxanthins; Trypan Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dye of lutein, zeaxanthin, trypan blue (Experimental): during the surgery will be evaluated if the dye is suitable for dyeing anterior lens capsule
  Interventions: Other: dye of lutein, zeaxanthin, trypan blue

INTERVENTIONS:
Other: dye of lutein, zeaxanthin, trypan blue — dye composed of lutein, zeaxanthin, trypan blue
  Other Names: combination of lutein, zeaxanthin, trypan blue

SUMMARY:
Effectiveness of lutein, zeaxanthin and trypan blue to stain the anterior lens capsule during cataract phacoemulsification.

DETAILED DESCRIPTION:
Twenty patients with cataract (nuclear, entumecente, total) and indication for cataract surgery will be selected to participate in this study.

ELIGIBILITY:
Inclusion Criteria

* Patients over 50 years
* Diagnosis of cataract (nuclear, entumecente, total)
* Absence of red reflex
* Indication of cataract surgery

Exclusion Criteria

* Posterior subcapsular cataract
* Any history of eye disease
* Glaucoma
* Eye infection affecting any structure prior ocular
* Any previous ocular surgery

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Visibility of the anterior lens capsule after the injection of dye | during the cataract surgery
  The visibility of the anterior lens capsule after the injection of dye, should be graduated as Bad OR Fair OR Good OR Fine

SECONDARY OUTCOMES:
Degree of impregnation of the dye | during the surgery
  The degree of impregnation of the anterior lens capsule by the dye should be graduated acording to the following scale:(0)not flushed; (1)stained weakly (light green); (2)moderately stained (medium green); (3)stained intensely (dark green)
usefulness of the dye | at the end of the cataract surgery
  the physician should evaluate the usufelness of the dye, according to the following scale: Bad, Fair, Good, Fine

CONTACTS AND LOCATIONS:
Overall Officials: Rubens Belfort Jr, MD, PhD, Principal Investigator — Fderal University of São Paulo
Locations (1):
- Dept. of Ophthalmology - UNIFESP/Hospital São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Vianna LM, Cohen MJ, Muccioli C, Lima A, Sousa-Martins D, Maia M, Belfort R Jr. Efficacy of a lutein-based dye (Phacodyne) for visualizing anterior capsulorhexis during cataract surgery by phacoemulsification. Arq Bras Oftalmol. 2014 May-Jun;77(3):173-7. doi: 10.5935/0004-2749.20140044. PMID 25295905